CLINICAL TRIAL: NCT00307320
Title: Coping With Stress During Pregnancy
Brief Title: Study Examining Stress During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 12234
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2008-08

CONDITIONS: Stress
Keywords: pregnancy; stress; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Relaxation Therapy

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Relaxation techniques
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: Relaxation Training — Relaxation techniques training
  Arms: 2

SUMMARY:
Researchers at UVa Health System are interested in how women experience and deal with stress during pregnancy. Participants will be randomly assigned either to engage in coping strategies on one's own or to receive 6 weeks of relaxation training. Researchers will examine how coping strategies affect the course of the pregnancy and the health of the infant

DETAILED DESCRIPTION:
Participants will be asked to fill out questionnaires and complete some tasks that require concentration as heart rate and other biological signals are monitored. Participants will also be asked to provide samples of saliva a few times during 1 day. These tasks will be repeated 3 times during pregnancy and participants will be asked to complete questionnaires at 6 months postpartum

A stress-reduction workshop will be offered to all participants at the completion of the study.

Participants will be paid for study completion

ELIGIBILITY:
Inclusion Criteria:

* beginning of the 2nd trimester of pregnancy
* feel stressed or overwhelmed
* do not yet have any children

Exclusion Criteria:

* more than 1 miscarriage
* currently receiving medication for anxiety or depression

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chambers, MA, Study Director — University of Virginia / University of Arizona; Susan Kirk, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Department of Psychology, Charlottesville, Virginia, United States